CLINICAL TRIAL: NCT03851120
Title: Promotion of Maternal Gut Microbiota and Psychological Stimulation on Child Cognitive Development at 6 Months of Age
Brief Title: Brain Probiotic and LC-PUFA Intervention for Optimum Early Life
Acronym: BRAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRAVE
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Maternal Exposure; Health Behavior; Infant Development; Child Development
MeSH Terms: conditions — Health Behavior | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Combination product: Probiotics and LC-PUFA The product will be given to 314 pregnant women, 157 pregnant women as an intervention group, and 157 pregnant women as a control group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator, and outcomes assessor do not know which one is the intervention product or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 150 pregnant women will be given Probiotics and 480 mg DHA, psychosocial stimulation, and healthy eating education
  Interventions: Dietary Supplement: Probiotics and LC-PUFA (480 mg DHA); Behavioral: Psychosocial stimulation and healthy eating education
- Control (Placebo Comparator): 150 pregnant women will be given placebo probiotics and 240 mg DHA, psychosocial stimulation, and healthy eating education
  Interventions: Dietary Supplement: Placebo probiotics and control LC-PUFA (120 mg DHA); Behavioral: Psychosocial stimulation and healthy eating education

INTERVENTIONS:
Dietary Supplement: Probiotics and LC-PUFA (480 mg DHA) — Probiotics and LC-PUFA (480 mg DHA)
  Arms: Intervention
Dietary Supplement: Placebo probiotics and control LC-PUFA (120 mg DHA) — Placebo probiotics and control LC-PUFA (120 mg DHA)
  Arms: Control
Behavioral: Psychosocial stimulation and healthy eating education — Psychosocial stimulation and healthy eating education

SUMMARY:
Probiotics is suggested to play several roles in promoting health, including alleviating disease symptoms, protection against atopic disease, and modulating the immune system by improving the beneficial gut microbiota colonization. The discovery of the gut microbiota-brain axis suggested that there is a reciprocal influence between the brain and the gut through a constant communication. This bi-directional axis enables signals to be transferred from brain to influence sensory, motor, and secretory modalities of the GI tract, also permits signal from the gut to influence brain function. The establishment of intestinal microbiota during early neurodevelopmental period suggests the colonization and maturation of gut microbiota may influence brain development. Several studies have shown there is an association between shifts in the gut microbiota composition in children with neurodevelopmental disorders. This study aims to investigate how maternal probiotic + LC-PUFA supported with government program supplements, healthy eating, and psychosocial stimulation could affect fetal brain development and later child brain functions and cognitive development. Intervention would be delivered to pregnant women for 9 months, starting at the end of second trimester of gestational period.

DETAILED DESCRIPTION:
Health and well-being at all ages is one of the goal set in the Sustainable Development Goals. Starting as early as possible has been considered to be an effective strategy for better investation in achieving healthy population. Therefore, the prevention and promotion of health and well being is starting to target population at younger age, starting as early as possible. Accordingly, the early life period of individuals has been considered as a critical period, especially in terms of the brain and cognitive development. The phases of brain development starts very early, starting from the fetal development in the uterus. The development process extends from early in the beginning of fetal development and lasted to the end, finishing last. The brain undergoes a period of rapid growth during the last trimester of fetal life and the first 2 years of childhood. Therefore, quality of pregnancy as well as quality of early life is important to the fetal brain development as well as later child brain function and cognitive development. In line with that notion, there are many studies suggesting that gut microbiota could affect CNS development through several ways, i.e. alteration of microbial composition, activation of immune system, changes in signaling via neural pathways, affecting tryptophan metabolism, modulating gut hormonal response and affecting hormonal signaling pathway, and releasing metabolites that could stimulate sympathetic nervous system. In particular, these studies have found bi-directional communication between the brain and the gut microbiota, referred to as the microbiota-gut-brain axis. The animal study showed that the gut microbiota regulates the development and function of the brain. Unfortunately, the study on human was still lacking.

This study is a randomized clinical trial (RCT) and placebo parallel controlled study, followed by a follow-up study at 2 years old. The research will be conducted in eight public hospitals / health care facilities in Indonesia, Jakarta.

In light of COVID-19 outbreak, if face-to-face activities are permitted by (1) national government (Indonesian Ministry of Health), (2) local government (DKI Jakarta), (3) the university, (4) Data Safety Monitoring Board, and (5) by consent of the subject, then the activities need to be strictly adjusted with the COVID-19 prevention measures for both personnel and subjects. All personnel and subjects who will be involved in the activities are required to fill out the COVID-19 symptom screening form prior to the visit.

Some adjustments for the project field implementation have been conducted during the outbreak, including:

1. Following Good Clinical Practice, for the safety of the subjects and all the team members, we are now ensuring that the subjects gain benefits from their involvement in the BRAVE project by implementing routine COVID-19 screening, providing adequate PPE for the fieldworkers, and educating them about the prevention measures.
2. Supplement delivery: Because we could not visit to the houses anymore due to staff restriction regulations, the bottles of the supplement are delivered using online motorcycle taxi services, and this includes the weighing scale for monthly monitoring. We have also developed a protocol to ensure the safety of supplement bottle transfer from the research personnel to the motorcycle taxi driver, and from the driver to the mothers, including safe distancing and disinfection procedures. We will also educate, provide a thermometer for self-temperature screening and provide the disinfectant to the mothers.
3. Outcome assessment: As per March 19, MRI assessment and blood sample collection remained implemented at a non-COVID-19 referral hospital and laboratory, with strict safety procedures for the subjects and personnel. For mothers who do not feel comfortable visiting the hospital/laboratory, they are free to refuse these procedures.
4. Compliance: Online system to promote and assess compliance. To maintain the quality, we cross-check mothers' activities by online assessment, interactive short message service (sms), and phone calls.
5. New Subject Recruitment are less priority right now or potentially stop for the time being until the situation is getting better.

ELIGIBILITY:
Inclusion Criteria:

Each pregnant woman must meet all of the following criteria to be enrolled in this study:

1. Indonesian pregnant women in the 2nd trimester of gestational period 2. healthy pregnancy (as measured by hemoglobin level, pregnancy status, pregnancy history) 3. Having a normal blood pressure 4. Planning to stay in the study area until the child is 6 months old 5. Willing to sign informed consent 5. Having a legally acceptable representative who is capable to understand the informed consent document and providing consent on the subject's behalf

Exclusion Criteria:

Each pregnant women meeting any of the following criteria will be excluded from the study:

1. Having foreign objects in the body due to trauma, artificial heart value, metal objects or ferromagnetic (plate, screw, clip, prosthetic), and electronic device (pacemaker, cochlear implant, insulin pump), and being claustrophobic
2. Having history of previous gestational diabetes or been diagnosed to have gestational diabetes
3. Having history of type 1 and type 2 diabetes
4. Severe anemia

Inclusion Criteria for Follow-up at 24 months:

1. Child age above 24 months from the BRAVE intervention project
2. Having a legally acceptable representative who is capable to understand the informed consent document and providing consent on the subject's behalf

Exclusion Criteria for Follow-up at 24 months:

1. Child being hospitalized during the study/data collection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 314 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Total brain volume | 1 year
  measured in parenchymal and cortical regions
Fetal brain development | 1 year
  Myelination index
Child cognitive at 4 months of age | 1 year
  Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III); a higher score indicates better performance
Brain function at 4 months of age | 1 year
  Brainstem Evoked Response Audiometry (BERA)
Eye tracking tasks at 6 months of age | 1 year
  Visual paired comparison memory task and Infant Orienting with Attention task at 4 months of age
Child cognitive at 6 months of age | 1 year
  Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III); a higher score indicates better performance

SECONDARY OUTCOMES:
Mother depression scale | 1 year
  Mother's Depression Test; a lower score indicates better performance
Birth weight | 4 month
  Baby weighing scale
Child's Growth | 6 months
  Change in weight-for-age z-score
Child's linear growth | 6 months
  Change in Length-for-age z-score
Head circumference | 6 months
  Change in Head-circumference-for-age
Child nutritional status | 6 months
  Change in weight-for-length z score
Quality of interaction with parents | 1 year
  Maternal involvement using HOME inventory questionnaires
Maternal blood micronutrient & macronutrient status | 1 year
  Zinc, iron, folate, omega-3 blood level
Incidence of gestational diabetes | 1 year
  Based on blood glucose assessment
Incidence of pre-eclampsia | 1 year
  Diagnosed by physician
Incidence of preterm birth | 4 month
  Gestational age
Mother's dietary quality | 1 year
  actual dietary intake, dietary pattern and quality
Maternal fecal microbiota composition | 1 year
  Microbiota composition by S16rRNA analysis
Child fecal microbiota composition | 4 months
  Microbiota composition by S16rRNA analysis
Maternal omega-3 level in breast milk at 4 months of age | 1 year
  Omega-3 level assessment using Gas Chromatography-Mass Spectrometry
Human milk oligosaccharides at 6 months of age | 1 year
  2-FL HMO assessment in breast milk
Maternal glucagon-like peptide-1 (GLP-1) profile | 1 year
  GLP-1 assessment using enzyme-linked immunosorbent assay
Maternal peptide-YY (PYY) profile | 1 year
  PYY assessment using enzyme-linked immunosorbent assay
Maternal fecal short chain fatty acids (SCFAs) | 1 year
  SCFAs analysis using Gas Chromatography-Mass Spectrometry
Child fecal short chain fatty acids | 1 year
  SCFAs analysis using Gas Chromatography-Mass Spectrometry
Post-partum weight retention | 1 year
  Monthly changes in maternal weight
Maternal weight circumference | 1 year
  Post-partum monthly changes in weight circumference
Gestational weight gain | 1 year
  Changes in maternal height throughout pregnancy period
Head circumference | 25 months
  Change in Head-circumference-for-age
Mid-Upper Arm Circumference | 25 months
  Change in Mid-Upper Arm Circumference
Toddler Body Weight | 25 months
  Toddler weighing scale
Toddler Height | 25 months
  Toddler height measurement
Mother Body weight | 1 year
  Mother's body weight
Mother Depression Test | 1 year
  Mother depression score
Mother Quality of Life | 1 year
  Mother quality of life score
Maternal History of COVID-19 during follow-up | 2 years
  Frequency of COVID-19 case during the follow-up period
Maternal Occurrence of COVID-19 during intervention period | 1 year
  Frequency of COVID-19 case during the intervention period
Child cognitive at 25-28 months of age | 1 year
  Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III); a higher score indicates better performance
Eye tracking tasks at 25-28 months of age | 1 year
  Visual paired comparison memory task and Infant Orienting with Attention task at 24 months of age
Mother Height | 1 year
  Mother's height
Mother Fat Percentage | 1 year
  Mother's fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, PhD, Principal Investigator — Human Nutrition Research Center, IMERI; Dep of Nutrition, Fac.of Medicine UI
Locations (1):
- Human Nutrition Research Center, Indonesian Medical Education Research Institute; and Department of Nutrition, Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
No plan to share Individual Participant Data (IPD) as stated in ClinicalTrial.gov registration. Data transfer to any third party will adhere to the ethical principles of the Declaration of Helsinki and comply with university regulations and the laws of the Republic of Indonesia, thereby upholding the rights of patients/subjects.

REFERENCES:
- [Background] Sheridan PO, Bindels LB, Saulnier DM, Reid G, Nova E, Holmgren K, O'Toole PW, Bunn J, Delzenne N, Scott KP. Can prebiotics and probiotics improve therapeutic outcomes for undernourished individuals? Gut Microbes. 2014 Jan-Feb;5(1):74-82. doi: 10.4161/gmic.27252. Epub 2013 Dec 16. PMID 24637591
- [Background] Sharon G, Sampson TR, Geschwind DH, Mazmanian SK. The Central Nervous System and the Gut Microbiome. Cell. 2016 Nov 3;167(4):915-932. doi: 10.1016/j.cell.2016.10.027. PMID 27814521
- [Background] Naaktgeboren, C. Effect of maternal probiotic exposure during pregnancy and lactation on the mother and infant. International Journal of Probiotics and Prebiotics 5: 113-124, 2010
- [Background] Ramakrishnan, U. A review of the benefits of nutrients supplements during pregnancy: from iron -folic-acid to long-chain polyunsaturated fatty acids to probiotics. Annales Nestle (English Ed): 29-40, 2010

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03851120/SAP_000.pdf